CLINICAL TRIAL: NCT03206931
Title: Expanded Access to Provide Selitrectinib (BAY2731954) for the Treatment of Cancers With a NTRK Gene Fusion.
Brief Title: Expanded Access to Provide Selitrectinib for the Treatment of Cancers With a NTRK Gene Fusion
Status: No longer available | Type: Expanded Access
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 21002
Record Dates: First submitted 2017-06-29; First posted 2017-07-02 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Solid Tumors Harboring NTRK Fusion
Keywords: Metastatic cancer; Advanced cancer; Neurotrophic tyrosine receptor kinase (NTRK); NTRK1; NTRK2; NTRK3; Fusion Positive; Children; Loxo-195
MeSH Terms: conditions — Neoplasm Metastasis | interventions — selitrectinib

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Selitrectinib (BAY2731954) — Selitrectinib is administered as capsules or liquid formulation.
  Other Names: Loxo-195

SUMMARY:
Selitrectinib expanded access is for minor and adult patients with cancer having a change in a particular gene (NTRK1, NTRK2, or NTRK3 gene fusion). The patients are ineligible for an ongoing selitrectinib clinical trial or have other considerations that prevent access to selitrectinib through an existing clinical trial. Expanded access is intended to treat individual patients with different types of cancers with a NTRK gene fusion, including blood cancers, who have previously received tropomyosin receptor kinase (TRK) inhibitor therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cancer with a NTRK1, NTRK2, and NTRK3 gene fusion
* Previous treatment with a kinase inhibitor with known activity on TRK inhibition
* Unable to participate in an ongoing selitrectinib clinical trial
* Medically suitable for treatment with selitrectinib

Exclusion Criteria:

* Currently enrolled in an ongoing clinical study with a TRK inhibitor

Min Age: 1 Month | Sex: All
Age Groups: Child, Adult, Older Adult